CLINICAL TRIAL: NCT00750451
Title: Empirical Low Molecular Weight Heparin Administration in the Luteal Phase in Patients With Recurrent Implantation Failures: a Randomized Open Labeled Trial
Brief Title: Low Molecular Weight Heparin in Recurrent Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AH-05/11
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Infertility; Fertilization in Vitro; Recurrent Implantation Failure
Keywords: fertilization in vitro; assisted reproduction; recurrent implantation failure; low molecular weight heparin; heparin; luteal phase
MeSH Terms: conditions — Infertility | interventions — Heparin, Low-Molecular-Weight; Crinone; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- LMWH (Experimental): Women in the LMWH arm are administered 1 mg/kg/day subcutaneously low molecular weight heparin after oocyte collection in addition to routine luteal phase support with vaginal progesterone
  Interventions: Drug: low molecular weight heparin (enoxaparine sodium)
- Control (Active Comparator): Women in the control arm are administered routine luteal phase support without the addition of LMWH
  Interventions: Drug: crinone 8% gel

INTERVENTIONS:
Drug: low molecular weight heparin (enoxaparine sodium) — 1 mg/kg/day subcutaneously in the luteal phase after IVF treatment
  Arms: LMWH
Drug: crinone 8% gel — routine luteal phase support with progesterone gel
  Arms: Control

SUMMARY:
Recurrent implantation failure is the failure to achieve a pregnancy after multiple attempts with in vitro fertilization treatment. The reason is usually obscure. Many empirical treatments have been offered without substantial evaluation. Heparin is thought to play a role in the embryo implantation process beyond its anticoagulation effects. The proposed study aims to assess the effectiveness and safety of empirical administration of low molecular weight heparin in patients undergoing a new IVF treatment cycle after multiple failed attempts.

ELIGIBILITY:
Inclusion Criteria:

* History of at least two previously failed fresh embryo transfer cycles
* All previously failed cycles to be performed in the American Hospital of Istanbul
* Female age ≤ 38 years
* Fresh ejaculate sperms to be used for ICSI
* No hormonal, coagulation, or immunological disorders detected
* Normal uterine cavity, as assessed by diagnostic office hysteroscopy or saline infusion sonography
* Normal female and male peripheral karyotype

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy beyond the 20th gestational week rate

SECONDARY OUTCOMES:
Clinical pregnancy rate
Embryo implantation rate

CONTACTS AND LOCATIONS:
Overall Officials: Cumhur B Urman, M.D., Study Director — American Hospital of Istanbul
Locations (1):
- Assisted Reproduction Unit of the American Hospital of Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Urman B, Ata B, Yakin K, Alatas C, Aksoy S, Mercan R, Balaban B. Luteal phase empirical low molecular weight heparin administration in patients with failed ICSI embryo transfer cycles: a randomized open-labeled pilot trial. Hum Reprod. 2009 Jul;24(7):1640-7. doi: 10.1093/humrep/dep086. Epub 2009 Apr 8. PMID 19357135